CLINICAL TRIAL: NCT03915639
Title: Effect of the Peri-incisional Multimodal Cocktail Infiltration on Postcraniotomy Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY 2018-035-01
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Pain, Postoperative
Keywords: Post-Craniotomy Headache; Postoperative Pain; Cocktail; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cocktail (Experimental): Participants in Group Cocktail are planned to infiltrate the head fixation sites after intubation and peri-incisionally prior to skin incision. The infiltration will be performed by the attending neurosurgeon. The muscle and the subcutaneous tissue beneath the fixation sites and incision site will be fully irrigated with the multimodal cocktail.
  Interventions: Procedure: Peri-incisional injection
- Ropivacaine (Active Comparator): Participants in Group Ropivacaine are planned to infiltrate the head fixation sites after intubation and peri-incisionally prior to skin incision. The infiltration will be performed by the attending neurosurgeon. The muscle and the subcutaneous tissue beneath the fixation sites and incision site will be fully irrigated with ropivacaine.
  Interventions: Procedure: Peri-incisional injection

INTERVENTIONS:
Procedure: Peri-incisional injection — The surgeons are planned to inject the cocktail mixture or ropivacaine to muscles and the subcutaneous tissue beneath the fixation sites and incision site using a 22-gauge needle in a sterile fashion prior to skin incision.

SUMMARY:
Postcraniotomy headache (PCH) has been underestimated for the past decades. However, current treatments for PCH are either considered insufficient or accompanied by severe side-effects. Some studies revealed that peri-incisional injection of a mixed cocktail that contains ropivacaine, epinephrine, ketorolac, and methylprednisolone showed significant efficacy in relieving postoperative pain after total hip or knee arthroplasty. Previous literature reported that the cause of PCH was related to incision of the scalp and dura, which is considered similar to causes to postoperative pain after total hip or knee arthroplasty. Thus, investigators suppose that the cocktail mixture can better relieve PCH in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Having signed the informed consent,
2. age 18-80 yrs,
3. American Society of Anaesthesiologists (ASA) physical status of I or II,
4. scheduled elective supratentorial craniotomy,
5. planned head fixation in a skull clamp.

Exclusion Criteria:

1. Allergy to LAs,
2. alcohol abuse,
3. intracranial hypertension,
4. active psychiatric disorders,
5. uncontrolled epilepsy,
6. chronic opioid use (more than 2 weeks),
7. undergoing a revision craniotomy,
8. high probability of having postoperative radio- or chemotherapy,
9. expectation of delayed extubation or no planned extubation,
10. pregnancy or breastfeeding during the study,
11. extreme body mass index (BMI) (less than 15 or more than 40),
12. preoperative Glasgow Coma Scale less than 15,
13. undergoing emergency or awake craniotomy surgery,
14. inability to understand the use of the NRS or the PCA. (Patients are informed of the instructions of NRS (from 0 to 10, where 0 and 10 represent no pain and the worst imaginable pain, respectively) and PCA after signing the informed consent the day before the operation. Patients who cannot understand the instruction of NRS and PCA will be excluded from the study.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative morphine consumption | 24 hours after recovery
  cumulative morphine consumption through PCA within 24 hours after recovery

SECONDARY OUTCOMES:
Postoperative 0-10 Numeric Rating Score | 1, 2, 4, 6, 12, 24, 48 and 72 hours after recovery and 3 and 6 months after craniotomy
  Numeric Rating Score is a common used scale in evaluating patients' pain intensity in clinical trials. The scale in the present trial is ranged from 0 to 10, where 0 represents no pain and 10 represents the worst imaginable pain. Higher values represent worse pain intensity.
Rate of post-operative opioid-related side effects | 1, 2, 4, 6, 12, 24, 48 and 72 hours after recovery
  Post-operative opioid-related side effects include post-operative opioid-induced oversedation, opioid-induced respiratory depression, pruritus, drowsiness, dizziness, blurred vision, and rash.
  Opioid-induced oversedation will be evaluated using the Pasero Opioid-induced Sedation Scale (POSS).
  1. Awake and alert,
  2. Slightly drowsy, easily aroused,
  3. Frequently drowsy, arousable, drift off to sleep during a conversation,
  4. Somnolent, minimal or no response to verbal or physical stimulation A POSS score of 3 or 4 is defined as oversedation.
  Opioid-induced respiratory depression (defined as respiratory rate <8/min and/or oxygen saturation <90% and/or apnoea ≥10 s, excessive sedation or upper airway obstruction.
Time interval to first PCA demand | within 24 hours after recovery
  The PCA device will automatically record the time interval to the first PCA demand based on a specially designed algorithm
Total PCA press counts | within 24 hours after recovery
  The PCA device will automatically record the total press counts based on a specially designed algorithm.
Total rescue medication usage | within 24 hours after recovery
  When PCA is not enough for analgesia, rescue medication will be used for relieving severe pain. The total rescue medication usage within 24 hours after recovery will be recorded.
Recovery | an average of 1 month
  Time to PACU discharge, time to ambulation, and length of stay (LOS)
Wound Healing Score | 3 and 6 weeks after craniotomy
  Wound Healing Score worksheet for assessment of outcomes in scalp clip versus artery forceps groups in patients undergoing craniotomy.
  The wound healing evaluation is based on skin healing, infection and hair regrowth.
  For skin healing, 1 represents fully healed, 2 represents ≤3 cm in total not healed, 3 represents >3 cm not healed, 4 represents areas of necrosis ≤3 cm, and 5 represents areas of necrosis >3 cm.
  For infection, 1 represents none, 2 represents ≤0.5-cm margin of redness , 3 represents more redness or superficial pus, 4 represents deep infection.
  For hair regrowth, 1 represents even regrowth along wound, 2 represents ≤3 cm not regrowing , 3 represents 3-6 cm not regrowing, 4 represents >6 cm not regrowing.
  Excellent wounds, total score of 3; Good wounds, Score 4-5; Suboptimal wounds, Score 6+
The size of surgical incision | at the end of the craniotomy
  Recording the size of surgical incision (unit: centimeter)
The duration of operation | at the end of the craniotomy
  Recording the duration of operation (unit:minute)
Rate of postoperative complications | within 30 days after craniotomy
  Postoperative complications include (1) Operative complications: intracranial infection, cerebral oedema, intracranial haematoma, CSF fistula, reoperation, reintubation and delayed extubation. incision infection, incision haematoma, delayed wound healing; (2) systemic complications: systemic infection, systemic inflammatory response syndrome and sepsis; (3) all-cause mortality
Postoperative antibiotic usage | within 30 days after craniotomy
  postoperative antibiotic usage

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rocha-Filho PA. Post-craniotomy headache: a clinical view with a focus on the persistent form. Headache. 2015 May;55(5):733-8. doi: 10.1111/head.12563. Epub 2015 Apr 22. PMID 25903913
- [Background] Papangelou A, Radzik BR, Smith T, Gottschalk A. A review of scalp blockade for cranial surgery. J Clin Anesth. 2013 Mar;25(2):150-9. doi: 10.1016/j.jclinane.2012.06.024. Epub 2013 Jan 23. PMID 23352875
- [Background] Akhigbe T, Zolnourian A. Use of regional scalp block for pain management after craniotomy: Review of literature and critical appraisal of evidence. J Clin Neurosci. 2017 Nov;45:44-47. doi: 10.1016/j.jocn.2017.08.027. Epub 2017 Sep 8. PMID 28890034
- [Background] Artime CA, Aijazi H, Zhang H, Syed T, Cai C, Gumbert SD, Ferrario L, Normand KC, Williams GW, Hagberg CA. Scheduled Intravenous Acetaminophen Improves Patient Satisfaction With Postcraniotomy Pain Management: A Prospective, Randomized, Placebo-controlled, Double-blind Study. J Neurosurg Anesthesiol. 2018 Jul;30(3):231-236. doi: 10.1097/ANA.0000000000000461. PMID 29117012
- [Background] Schankin CJ, Gall C, Straube A. Headache syndromes after acoustic neuroma surgery and their implications for quality of life. Cephalalgia. 2009 Jul;29(7):760-71. doi: 10.1111/j.1468-2982.2008.01790.x. Epub 2009 Feb 23. PMID 19239675
- [Background] Flexman AM, Ng JL, Gelb AW. Acute and chronic pain following craniotomy. Curr Opin Anaesthesiol. 2010 Oct;23(5):551-7. doi: 10.1097/ACO.0b013e32833e15b9. PMID 20717011
- [Background] Kerr DR, Kohan L. Local infiltration analgesia: a technique for the control of acute postoperative pain following knee and hip surgery: a case study of 325 patients. Acta Orthop. 2008 Apr;79(2):174-83. doi: 10.1080/17453670710014950. PMID 18484242
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Parvataneni HK, Shah VP, Howard H, Cole N, Ranawat AS, Ranawat CS. Controlling pain after total hip and knee arthroplasty using a multimodal protocol with local periarticular injections: a prospective randomized study. J Arthroplasty. 2007 Sep;22(6 Suppl 2):33-8. doi: 10.1016/j.arth.2007.03.034. Epub 2007 Jul 26. PMID 17823012
- [Background] Lamplot JD, Wagner ER, Manning DW. Multimodal pain management in total knee arthroplasty: a prospective randomized controlled trial. J Arthroplasty. 2014 Feb;29(2):329-34. doi: 10.1016/j.arth.2013.06.005. Epub 2013 Jul 11. PMID 23850410
- [Background] Milani P, Castelli P, Sola M, Invernizzi M, Massazza G, Cisari C. Multimodal Analgesia in Total Knee Arthroplasty: A Randomized, Double-Blind, Controlled Trial on Additional Efficacy of Periarticular Anesthesia. J Arthroplasty. 2015 Nov;30(11):2038-42. doi: 10.1016/j.arth.2015.05.035. Epub 2015 May 23. PMID 26072302
- [Background] Spangehl MJ, Clarke HD, Hentz JG, Misra L, Blocher JL, Seamans DP. The Chitranjan Ranawat Award: Periarticular injections and femoral & sciatic blocks provide similar pain relief after TKA: a randomized clinical trial. Clin Orthop Relat Res. 2015 Jan;473(1):45-53. doi: 10.1007/s11999-014-3603-0. PMID 24706022
- [Background] Vendittoli PA, Makinen P, Drolet P, Lavigne M, Fallaha M, Guertin MC, Varin F. A multimodal analgesia protocol for total knee arthroplasty. A randomized, controlled study. J Bone Joint Surg Am. 2006 Feb;88(2):282-9. doi: 10.2106/JBJS.E.00173. PMID 16452738